CLINICAL TRIAL: NCT03007069
Title: Implant Insertion in Defective Anterior Maxillary Ridge Augmented Using Mineralized Plasmatic Matrix Versus Autogenous Bone Graft
Brief Title: Preimplant Site Augmentation Using MPM Versus Autogenous Bone Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Usama Mahmoud El Masry, Dentist at menistry of health, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CairoMPM-ABG
Record Dates: First submitted 2016-12-25; First posted 2017-01-02 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-12

CONDITIONS: Bone Resorption
MeSH Terms: conditions — Bone Resorption | interventions — 1-methyl-1-piperidinomethane sulfonate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autogenous bone graft (Gold Standard). (Experimental): Patients with defective maxillary alveolar ridges requiring implant insertion will have Autogenous bone graft (Gold standard) and collagen membrane to be used for bone augmentation around exposed threads of inserted dental implants.
  Interventions: Other: Autogenous bone graft (gold standard).
- MPM Augmentation. (Active Comparator): Mineralized plasmatic matrix (MPM) to be used without collagen membrane to augment the defect in the maxillary bone and cover the exposed threads of the dental implants.
  Interventions: Other: Mineralized plasmatic matrix (MPM).

INTERVENTIONS:
Other: Mineralized plasmatic matrix (MPM). — By using venoud blood from the patient, together with bone graft, a centrifuge will be used to obtain the top layer after centrifuging blood at 3000 RPM, for 10 minutes , Which will result if sticky bone graft consistency after mixing.
  Other Names: Sticky bone graft.
  Arms: MPM Augmentation.
Other: Autogenous bone graft (gold standard). — Exposed implant threads are to be covered with autogenous bone and collagen membrane.
  Other Names: Autobone.
  Arms: Autogenous bone graft (Gold Standard).

SUMMARY:
Using growth factors obtained from patient's venous blood mixed with particulate autogenous bone the study compares bone gain by implant with gold standards.

DETAILED DESCRIPTION:
To study the effectiveness of MPM in ridge augmentation with implant insertion compared with autogenous bone graft.

-PICO-

Population (P): Patients with defective maxillary alveolar ridge requiring implant insertion.

Intervention (I): Ridge augmentation with MPM.

Comparator (C): Autogenous bone graft.

Outcome (O): Patient satisfaction - Implant stability.

ELIGIBILITY:
Inclusion Criteria:

1. Medically free patients.
2. Evaluated bone height on CBCT to be (0-4 mm buccal bone dehiscence) and width (not less than 4.5 mm)
3. Patients with Anterior maxillary defective partially edentulous ridge.
4. Age between 18 and 40 years.
5. Both sexes.
6. Patients physically able to tolerate surgical and restorative procedures.
7. Patients with an opposing tooth to the pre-implant site.
8. Good oral hygiene.
9. Highly motivated patients.

Exclusion Criteria:

1. Patients allergic to local anesthetic agent.
2. Pregnant or lactating females.
3. Presence of any pathosis in the pre-implant site.
4. Presence of any mucosal disease.
5. Presence of parafunctional habits.
6. History of oral radiotherapy.
7. History of prolonged steroids use.
8. Psychological disorders.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction regarding esthetic results , outcome will be measure using questionnaire. | 5 months

SECONDARY OUTCOMES:
Stability of dental implants , this will be measured using Ostell device in ISQ units. | 5 months.

IPD SHARING:
Plan to Share IPD: No
Evaluation of the comparative Effectiveness of MPM Augmentation in Anterior ridge defects with Autogenous bone graft.